CLINICAL TRIAL: NCT04927702
Title: Assessment of Wound Closure Comparing Synthetic Hybrid-Scale Fiber Matrix With Standard of Care in Treating Diabetic Foot Ulcers (DFU) and With Living Cellular Skin Substitute in Treating Venous Leg Ulcers (VLU)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to slow enrollment
Sponsor: Acera Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-RES-001
Record Dates: First submitted 2021-06-03; First posted 2021-06-16 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Diabetic Foot Ulcer Participants Assigned to Synthetic Hybrid-Scale Fiber Matrix (Restrata®) (Experimental): Biweekly (every 2 weeks) application for either 12 weeks or until 100 percent epithelialization / wound closure (whichever occurs first)
  Interventions: Device: Synthetic Hybrid-Scale Fiber Matrix
- Diabetic Foot Ulcer Participants Assigned to Standard of Care (Active Comparator): Weekly application for either 12 weeks or until 100 percent epithelialization / wound closure (whichever occurs first)
  Interventions: Device: Standard of Care
- Venous Leg Ulcer Participants Assigned to Synthetic Hybrid-Scale Fiber Matrix (Restrata®) (Experimental): Biweekly (every 2 weeks) application for either 16 weeks or until 100 percent epithelialization / wound closure (whichever occurs first)
  Interventions: Device: Synthetic Hybrid-Scale Fiber Matrix
- Venous Leg Ulcer Participants Assigned to Living Cellular Skin Substitute (Apligraf®) (Active Comparator): Biweekly (every 2 weeks) application for either 16 weeks or until 100 percent epithelialization / wound closure (whichever occurs first)
  Interventions: Device: Living Cellular Skin Substitute

INTERVENTIONS:
Device: Synthetic Hybrid-Scale Fiber Matrix — A synthetic absorbable skin substitute indicated for use in the local management of wounds. It is made of small synthetic fibers that are designed to be similar to the structure of human skin.
  Other Names: Restrata
  Arms: Diabetic Foot Ulcer Participants Assigned to Synthetic Hybrid-Scale Fiber Matrix (Restrata®); Venous Leg Ulcer Participants Assigned to Synthetic Hybrid-Scale Fiber Matrix (Restrata®)
Device: Standard of Care — To ensure off-loading, each patient will be fitted with an off-loading device based on the investigator's decision, e.g. a boot for forefoot and a heel protector for hindfoot. Patients is instructed on how to care for the surgical site, utilize an off-loading device, and keep the surgical site moist and clean. If the wound is dry, a hydrogel category dressing type should be used. If the wound has exudate, an alginate or foam dressing is recommended.
  Arms: Diabetic Foot Ulcer Participants Assigned to Standard of Care
Device: Living Cellular Skin Substitute — An absorbable skin substitute comprised of human and bovine (cow) tissues indicated for use in the local management of wounds.
  Other Names: Apligraf
  Arms: Venous Leg Ulcer Participants Assigned to Living Cellular Skin Substitute (Apligraf®)

SUMMARY:
In participants with diabetic foot ulcers (DFUs), this study will assess complete wound closure by comparing synthetic hybrid-scale fiber matrix (Restrata®) with standard of care.

In participants with venous leg ulcers (VLUs), this study will assess complete wound closure by comparing synthetic hybrid-scale fiber matrix (Restrata®) with living cellular skin substitute (Apligraf®)

ELIGIBILITY:
Inclusion Criteria for Participants with Diabetic Foot Ulcers:

1. Participant is at least 18 years old
2. Participant is willing and capable of complying with all protocol requirements
3. Participant or legally authorized representative (LAR) is willing to provide written informed consent
4. Participant has Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per American Diabetes Association)
5. Ulcer(s) must be located at least in part on the foot or ankle
6. Ulcer(s) must be present for more than 28 days prior to randomization and initial application of study product, and has not adequately responded to conventional ulcer therapy
7. Wound size must be >1.0 cm^2 and < 25 cm^2 on the day of randomization and initial application of the study product, after initial debridement
8. Participant has adequate circulation to the affected extremity(ies), as demonstrated by at least ONE of the following within 60 days prior to enrollment/randomization:

   1. Dorsum transcutaneous oxygen test (TcPO2) of study leg(s) with results ≥40mmHg, OR
   2. Ankle-Brachial Index (ABI) of study leg(s) with results of ≥ 0.7 and ≤ 1.3, OR
   3. Toe-Brachial Index (TBI) of study extremity(ies) with results of ≥ 0.5

Exclusion Criteria for Participants with Diabetic Foot Ulcers:

1. Participant has been previously enrolled into this study, or is currently participating in another prospective drug or device study that has not reached its primary endpoint
2. Participant is pregnant, breast feeding or planning to become pregnant
3. Participant has a known allergy to resorbable suture materials, e.g. Polyglactin 910 (PGLA), Polydioxanone (PDS)
4. Participant has a life expectancy less than six months as assessed by the investigator
5. Participant has received skin substitutes during the screening period or within 14 days prior to beginning of screening period
6. Participant has an additional wound within 3 cm of the study wound(s) or study wounds are less than 3 cm apart
7. Hgb A1c > 12 percent within 3 months prior to randomization
8. Participant not in reasonable metabolic control in the judgment of the investigator
9. Participant with a known history of poor compliance with medical treatments
10. Participant currently undergoing cancer treatment
11. Participant has been diagnosed with at least one of the following autoimmune connective tissue diseases: lupus, vasculitis, sickle cell, or uncontrolled rheumatoid arthritis
12. Participant is taking parenteral corticosteroids or any cytotoxic agents for 7 consecutive days during the screening period or up to 30 days before the screening period. Chronic oral steroid use is not excluded if dose is < 10 mg per day for prednisone.
13. Active infection, undrained abscess, or critical colonization of the wound(s) with bacteria in the judgment of the investigator
14. Osteomyelitis or exposed bone, probes to bone or joint capsule on investigator's exam or radiographic evidence
15. Participant unwilling or unable to safely utilize appropriate offloading device to unweight wound(s)
16. Study ulcer(s) experiences greater than 30 percent reduction over the 2-week screening period
17. Participant also has a venous leg ulcer that is enrolled into this study

Inclusion Criteria for Participants with Venous Leg Ulcers:

1. Participant is at least 18 years old
2. Participant is willing and capable of complying with all protocol requirements
3. Participant or legally authorized representative (LAR) is willing to provide written informed consent
4. Participant has peripheral venous disease per investigator judgment or diagnostic confirmation
5. Ulcer(s) must be venous in origin, located on a lower extremity
6. Ulcer(s) must be present for more than 28 days prior to randomization and initial application of study product, and has not adequately responded to conventional ulcer therapy
7. Wound(s) size must be >1.0 cm^2 and < 50 cm^2 on the day of randomization and initial application of the study product, after initial debridement
8. Participant has adequate circulation to the affected extremity(ies), as demonstrated by at least ONE of the following within 60 days prior to enrollment/randomization:

   1. Dorsum transcutaneous oxygen test (TcPO2) of study leg(s) with results ≥ 40mmHg, OR
   2. Ankle-brachial index (ABI) of study leg(s) with results of ≥ 0.7 and ≤ 1.52, OR
   3. Toe-Brachial Index (TBI) of study leg(s) with results of ≥ 0.5, OR
   4. Doppler arterial waveforms, which are triphasic or biphasic at the ankle of the affected leg(s)

Exclusion Criteria for Participants with Venous Leg Ulcers:

1. Participant has been previously enrolled into this study, or is currently participating in another prospective drug or device study that has not reached its primary endpoint
2. Participant is pregnant, breast feeding or planning to become pregnant
3. Participant has a known allergy to resorbable suture materials, e.g. Polyglactin 910 (PGLA), Polydioxanone (PDS)
4. Participant has a known allergy to bovine materials or agarose shipping materials
5. Participant has a life expectancy less than six months as assessed by the investigator
6. Participant has received skin substitutes during the screening period or within 14 days prior to the beginning of the screening period
7. Participant has an additional wound within 3 cm of the study wound or study wounds are less than 3 cm apart
8. Hgb A1c > 12 percent within 3 months prior to randomization in patients with a known history of diabetes
9. Participant is not in reasonable metabolic control in the judgment of the investigator
10. Participant has a known history of poor compliance with medical treatments
11. Participant currently undergoing cancer treatment
12. Participant has been diagnosed with at least one of the following autoimmune connective tissue diseases: lupus, vasculitis, sickle cell, or uncontrolled rheumatoid arthritis
13. Participant is taking parenteral corticosteroids or any cytotoxic agents for 7 consecutive days during the screening period or up to 30 days before the screening period. Chronic oral steroid use is not excluded if dose is < 10 mg per day for prednisone.
14. Active infection, undrained abscess, or critical colonization of the wound(s) with bacteria in the judgment of the investigator
15. Participant unwilling or unable to tolerate use of compression therapy for the duration of the study
16. Study ulcer(s) experiences greater than 30 percent reduction over the 2-week run-in period
17. Participant also has a diabetic foot ulcer that is enrolled into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
For Participants With Diabetic Foot Ulcers, number of participants with 100 Percent Epithelialization (Closure) of Wound | 12 weeks
  100 percent epithelialization of wound as assessed by a blinded evaluator via review of a three-dimensional high resolution photo of the wound plus confirmation of no drainage or need for additional dressing 2 weeks after 100 percent epithelialization
For Participants With Venous Leg Ulcers, number of participants with 100 Percent Epithelialization (Closure) of Wound | 16 weeks
  100 percent epithelialization of wound as assessed by a blinded evaluator via review of a three-dimensional high resolution photo of the wound plus confirmation of no drainage or need for additional dressing 2 weeks after 100 percent epithelialization

SECONDARY OUTCOMES:
Decrease in Wound Area | Weekly assessments for 12 weeks for DFU participants (16 weeks for VLU participants), or until 100 percent epithelialization, whichever occurs first.
  Wound area measurements will be made via a three-dimensional high resolution photo of the wound with automated measurements.
Time to 100 Percent Epithelialization | 12 weeks for DFU participants (16 weeks for VLU participants), or until 100 percent epithelialization, whichever occurs first.
  The number of weeks from initial application of study product until 100 percent epithelialization is first identified.
Number of Product Applications | 12 weeks for DFU participants (16 weeks for VLU participants), or until 100 percent epithelialization, whichever occurs first
  The number of applications of study product until 100 percent epithelialization is first identified

OTHER OUTCOMES:
Score on SF-36 Questionnaire Measuring Quality of Life | Day of initial product application and at either 12 weeks for DFU participants (16 weeks for VLU participants) or at 100 percent epithelialization (whichever occurs first)
Pain Reported By Participant | Day of initial product application and at either 12 weeks for DFU participants (16 weeks for VLU participants) or at 100 percent epithelialization (whichever occurs first)
  The pain reported by the participant on a scale of 0 through 10 with 10 being the highest level of pain the participant has experienced
Number of Adverse Events Related to the Study Product and/or Procedure | Up to six months
Investigator's Rating of the Ease of Use and Handling of Study Product | 12 weeks for DFU participants (16 weeks for VLU participants), or until 100 percent epithelialization, whichever occurs first
  Investigator's rating of the ease of use and handling of the study product. Investigator will rate study product as "very satisfied", "satisfied", or "not satisfied"
Cost Effectiveness | 12 weeks for DFU participants (16 weeks for VLU participants), or until 100 percent epithelialization, whichever occurs first
  Total cost of study product applied to the participant
Number of participants with coverage of product by payor (insurance) | 12 weeks for DFU participants (16 weeks for VLU participants), or until 100 percent epithelialization, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - ILD Research Center, Vista, California
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Barry University, Miami Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Gundersen Health System, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No